CLINICAL TRIAL: NCT06031324
Title: The Role of Lung Ultrasonography Score in Predicting Prognosis in Term and Late Preterm Newborns With Postnatal Respiratory Distress
Acronym: TeLaPLUS
Status: Recruiting | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Bayram Ali DORUM, Associate Professor of Neonatology, Bursa City Hospital
Other Study IDs: BCH-2023-14/2
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Distress Syndrome; Lung Ultrasonography Score
Keywords: Respiratory distress syndrome; Lung ultrasonography; Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory distress in term and late preterm infants in the first hour after birth is a prevalent condition. This situation may occur due to different reasons such as minimal respiratory stress, transient tachypnea of newborn, respiratory distress syndrome, and congenital pneumonia. It can be not easy to distinguish this in the first hours. This study aimed to investigate the place of the lung ultrasonography score in the prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Having symptoms of respiratory distress that begin soon after birth,
* > 34 gestational age,
* >1900 gr birth weight,
* Family consent

Exclusion Criteria:

* Congenital anomaly
* Chromosomal anomaly
* Hydrops fetalis
* Congenital heart disease

Ages: 30 Minutes to 120 Minutes | Sex: All
Age Groups: Child
Study Population: Term and late-preterm premature newborns with respiratory distress symptoms in the first 30 minutes after birth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Enrollment of a targeted number of patients | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)